CLINICAL TRIAL: NCT04246697
Title: Multimodal Management for Perioperative Analgesia in Otolaryngology - Head and Neck Free Flap Reconstructive Surgery: A Prospective Study
Brief Title: Multimodal Pain Study in Free Flap Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00025711
Record Dates: First submitted 2019-10-31; First posted 2020-01-29 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Cancer; Analgesia
MeSH Terms: conditions — Head and Neck Neoplasms; Agnosia | interventions — Acetaminophen; Oxycodone; Morphine; Gabapentin; Ketorolac Tromethamine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care A (Active Comparator): Randomized controlled prospective trial to compare two standards of care for head and neck surgery pain management. Arm A, will include:
  * Scheduled Tylenol 1000 mg IV one time dose intra-operatively, then 650 mg via PEG tube or PO Q4H to a max dose of 4gm/24 hrs
  * Opioids prn based on Numeric Pain Scale (0-10, with 0 indicating no pain and 10 indicating worst pain ever):
  * 0-3: no prn meds, reassurance, listen to music, watch TV.
  * 4-7: Oxycodone 5 mg q4h prn via PEG tube or PO with a maximum of 30 mg/24 hours.
  * 8-10 Morphine 2 mg IV q2h prn breakthrough pain.
  Interventions: Drug: Tylenol; Drug: Oxycodone; Drug: Morphine
- Standard of Care B (Experimental): Arm B, will include:
  * Arm A description with addition..
  * Scheduled Ketorolac starting post-op day #1, 15 mg q6h (max 120 mg/day), for a total of 5 days
  * Scheduled Gabapentin starting 7 days preoperatively to continue postoperatively
  * Regional block per anesthesia protocol - Initial block: 0.5% bupivacaine, 20 ml Continuous infusion: 0.125% bupivacaine at 6 ml/hr with a 5 ml bolus available every 30 mins
  Interventions: Drug: Tylenol; Drug: Oxycodone; Drug: Morphine; Drug: Gabapentin; Drug: toradol; Drug: Bupivacaine

INTERVENTIONS:
Drug: Tylenol — Used for both arms, scheduled
Drug: Oxycodone — Used for both arms PRN
Drug: Morphine — Used for both arms PRN
Drug: Gabapentin — Used for Arm B
  Arms: Standard of Care B
Drug: toradol — Used for Arm B
  Arms: Standard of Care B
Drug: Bupivacaine — Used for Arm B - anesthesia block
  Arms: Standard of Care B

SUMMARY:
This study will be fashioned as a randomized, prospective study comparing Pain Management Arm A and Pain Management Arm B. Arm A will have scheduled Tylenol with opioids available as needed (PRN) in the peri-operative period. Arm B will undergo scheduled Gabapentin, Ketorolac and Tylenol as well as the Anesthesiology team managing regional nerve blocks, with opioids available PRN in the peri-operative period. The amount of pain medication used by all patients will be recorded as well as pain scores documented on a pain scale (0-10 with 0 indicating no pain and 10 indicating worst pain ever) as well as ABC pain scale throughout the patients' hospital stay. Morphine equivalents for the opioids will be calculated for each arm while observing pain scores. Then, the investigators will compare these two groups to see if there is a difference in opioid pain medication used. The study team's hypothesis is that the use of Gabapentin, Ketorolac, and Tylenol in combination will significantly reduce (at least 30% of Mean Morphine Equivalents - MME) the use of opioid medication for patients undergoing head and neck free flap reconstruction with similar to improved pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who are seen in the Department of Otolaryngology-Head and Neck Surgery clinic.
* Patients with a new H&N cancer diagnosis undergoing primary surgery (free flap) for their cancer treatment.

Exclusion Criteria:

* Prior treatment for head and neck cancer.
* Planned treatment with primary radiation or chemoradiation for their head and neck cancer.
* Pregnant or lactating women.
* Patients with a history of consistent or regular opioid use for greater than six months used pre-operatively.
* Chronic gabapentin, pregabalin, and other non-opioid pain medication use pre-operatively.
* Diagnoses with fibromyalgia, anxiety disorder and other pain syndromes.
* Patients with documented history of kidney or liver disease.
* Patients with pre-operative lab values concerning for kidney/liver disease such as increased creatinine or liver function tests.
* Patients with a history of a serious GI bleed, CAD, or history of ischemic stroke .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Mean morphine equivalents for Arm A | During the study period of approximately 1 year
  Mean morphine equivalents will be calculated after converting all opioids to morphine equivalents and then averaging them.
Mean morphine equivalents for Arm B | During the study period of approximately 1 year
  Mean morphine equivalents will be calculated after converting all opioids to morphine equivalents and then averaging them.

SECONDARY OUTCOMES:
Length of stay | Analyze the first 7 post-operative days but take note of how long they stayed.
  Length of stay in days
Post-operative complications | Analyze the first 7 post-operative days
  Monitor chart/EMR for bleeding, acute kidney injury, etc.
Pain assessment for patients | Nurses will use the DVPRS for each assessment while the patient is hospitalized, typically for seven days. Nursing assessments typically are Q2H-Q4H.
  Pain assessment will occur with nurses providing patient a 0-10 pain scale (i.e. 0 being the lowest and 10 being the greatest amount of pain) named the Defense Veterans Pain Rating Scale for each nursing assessment in order to know which pain medications to administer.
Pain assessment for patients | The ABC pain scale will be given once daily for the patient to fill out for the first seven days.
  There is another pain assessment scale that will be distributed once daily to the patients to assess their pain and how it is affecting their functionality. This pain assessment/survey is named the ABC pain scale, which is a qualitative pain assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Shnayder, MD, Principal Investigator — KUMC
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided